CLINICAL TRIAL: NCT04819776
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Iloperidone for 4 Weeks in the Treatment of Patients With Acute Manic Episodes Associated With Bipolar I Disorder
Brief Title: Evaluation of Efficacy and Safety of Iloperidone in the Acute Treatment of Manic or Mixed Episodes Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VYV-683-3201
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — iloperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iloperidone (Experimental)
  Interventions: Drug: Iloperidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Iloperidone Placebo

INTERVENTIONS:
Drug: Iloperidone — Oral iloperidone
  Other Names: FANAPT®; VYV-683
  Arms: Iloperidone
Drug: Iloperidone Placebo — Oral placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the efficacy, safety, and tolerability of iloperidone compared with placebo in treating acute manic or mixed episodes associated with Bipolar I Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 to 65 years of age (inclusive)
* Diagnosed with bipolar I disorder, manic or mixed-type, per DSM-5 criteria
* Voluntary hospitalization for current manic episode

Exclusion Criteria:

* Patients with a DSM-5 diagnosis of a psychiatric disorder other than bipolar I disorder that was the primary focus of treatment within the previous six months
* Patients who are experiencing a first manic episode or meeting criteria for rapid cycling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (20):
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Rogers, Arkansas
  - Vanda Investigational Site, Cerritos, California
  - Vanda Investigational Site, Culver City, California
  - Vanda Investigational Site, Long Beach, California
  - Vanda Investigational Site, Orange, California
  - Vanda Investigational Site, Torrance, California
  - Vanda Investigational Site, Miami Lakes, Florida
  - Vanda Investigational Site, Oakland Park, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Decatur, Georgia
  - Vanda Investigational Site, Gaithersburg, Maryland
  - Vanda Investigational Site, Flowood, Mississippi
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Marlton, New Jersey
  - Vanda Investigational Site, Dayton, Ohio
  - Vanda Investigational Site, North Canton, Ohio
  - Vanda Investigational Site, Austin, Texas
  - Vanda Investigational Site, DeSoto, Texas
  - Vanda Investigational Site, Richardson, Texas
- Bulgaria (6):
  - Vanda Investigational Site, Novi Iskar, Sofia-Grad
  - Vanda Investigational Site, Tserova Koria, Veliko Tarnovo
  - Vanda Investigational Site, Kardzhali
  - Vanda Investigational Site, Lovech
  - Vanda Investigational Site, Veliko Tarnovo
  - Vanda Investigational Site, Vratsa
- Vanda Investigational Site, Tuszyn, Poland

REFERENCES:
- [Derived] Torres R, Czeisler EL, Chadwick SR, Stahl SM, Smieszek SP, Xiao C, Polymeropoulos CM, Birznieks G, Polymeropoulos MH. Efficacy and Safety of Iloperidone in Bipolar Mania: A Double-Blind, Placebo-Controlled Study. J Clin Psychiatry. 2024 Jan 15;85(1):23m14966. doi: 10.4088/JCP.23m14966. PMID 38236020

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety analyses included patients who received 1 or more doses of study medication. Of the 417 randomized, 414 received at least one dose of study medication.
Period: Overall Study
Arm/Group | Iloperidone | Placebo
Started | 206 | 208
Completed | 139 | 153
Not Completed | 67 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloperidone | Placebo | Total
Number analyzed (Participants) | 206 | 208 | 414
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (12.76) | 43.9 (12.55) | 43.4 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 96 | 186
  Male | 116 | 112 | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 133 | 132 | 265
  Black or African American | 62 | 55 | 117
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 3 | 4
  Other | 9 | 15 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Young Mania Rating Scale (YMRS) Total Score
Description: The Young Mania Rating Scale (YMRS) is an 11-item scale. Individual item scores are summed for a total possible score of 0 (best) to 60 (worst).
Time Frame: Week 4
Population: Efficacy analyses were based on the Intent-To-Treat (ITT) population, which included all randomized patients who received a dose of study drug and had at least one valid post-baseline efficacy measurement while on study medication. Of the 417 randomized, 392 received at least one dose of study medication and had at least one valid post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: Change from Baseline in YMRS Total Score
Arm/Group | Iloperidone | Placebo
Number analyzed (Participants) | 198 | 194
Change from Baseline in YMRS Total Score | -14.0 (0.64) | -10.0 (0.63)

ADVERSE EVENTS:
Time Frame: AE data was collected during the 28 day study period plus a 7 day follow up period.
Arm/Group | Iloperidone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/208
Serious Adverse Events (participants affected / at risk) | 4/206 | 1/208
Other Adverse Events (participants affected / at risk) | 88/206 | 25/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone (N=206) | Placebo (N=208)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bipolar disorder (depression) (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone (N=206) | Placebo (N=208)
Tachycardia (Cardiac disorders) | 36 | 11
Dizziness (Nervous system disorders) | 23 | 2
Dry mouth (Gastrointestinal disorders) | 19 | 4
Alanine aminotransferase increased (Investigations) | 15 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Weight increased (Investigations) | 12 | 3
Somnolence (Nervous system disorders) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT04819776/Prot_SAP_000.pdf